CLINICAL TRIAL: NCT03743207
Title: Preterm Infants May Better Tolerate Feeds at Temperatures Closer to Freshly Expressed Breast Milk- A Randomized Controlled Trial
Brief Title: Preterm Infants May Better Tolerate Warmer Feeds
Acronym: Prematurity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Ozge Altun Koroglu, Associated Professor, M.D., Ege University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: EGE20121284
Record Dates: First submitted 2018-10-30; First posted 2018-11-16 (Actual); Last update posted 2018-11-16 (Actual); Status verified 2018-11

CONDITIONS: Prematurity; Feeding Disorder Neonatal
Keywords: Prematurity; Enteral nutrition; Feeding tolerance; Temperature
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The infants were randomly assigned using the last digit of their hospital identification number to two different groups with different feeding temperatures. Only the nurse giving the primary care was not blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Room temperature (Experimental): All of the infants in neonatal intensive care units are used to be fed with milk at 22-24°C which is close to room temperature.
  Interventions: Other: Room temperature
- Warmer temperature (Experimental): The investigators decided to feed the infants in this group with warmer milk at to examine the effects of feeding temperature.
  Interventions: Other: Warmer temperature

INTERVENTIONS:
Other: Room temperature — These infants were fed with room temperature (22-24 °C) so that hypothesizing that they will have more feeding tolerance and therefore more co-existing morbidities.
  Arms: Room temperature
Other: Warmer temperature — Fifteen NICU mothers volunteered and expressed their milk for rapid measurement of freshly expressed breast milk. The mean (± SD) temperature of freshly expressed breast milk was found to be 33±1.5 °C in these preliminary measurements. Confirming this finding, the investigators decided to feed these infants with milk at 32 - 34 °C to examine the effects of feeding temperature and the possible comorbidities with a hypothesis that warmer feeding at the temperature of freshly expressed breast milk may be better physiologically.
  Arms: Warmer temperature

SUMMARY:
Feeding intolerance is frequent among preterm infants in neonatal intensive care units (NICUs). Although there are many studies about enteral nutrition strategies and content in preterm infants, no evidence-based standards exist for the optimal milk temperature for preterm infants. Therefore, in this study the investigators aimed to examine the effects of feeding temperature and the possible morbidities.

DETAILED DESCRIPTION:
Feeding intolerance is one of the most frequent problems among preterm infants. These infants are fed with expressed breast milk or preterm formulas of which the temperature is not routinely measured. In this study, the investigators aimed to examine the effects of feeds with warm versus room temperature milk in preterm infants. Infants with a birth weight of ≤1500 g or gestational age of ≤ 34 weeks were included in the study and assigned to two different feeding temperature groups (22-24°C and 32-34°C). Some infants in both groups were exclusive breast milk fed and some received artificial milk. Feeding tolerance of patients in both groups and the consequences were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Infants born to birth weight of ≤1500 g
* Infants born to gestational age of ≤ 34 weeks

Exclusion Criteria:

* Genetic syndrome
* Gastrointestinal system anomalies
* Patients born small for their gestational age

Ages: 1 Day to 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2012-10-01 (Actual); Primary Completion 2014-04-30 (Actual); Study Completion 2014-04-30 (Actual)

PRIMARY OUTCOMES:
Gastric residual volume in mililitres after every feeding | through study completion, an average of 6 months
  Gastric residual volume amount during the study

SECONDARY OUTCOMES:
Transition time to total enteral feeding | through study completion, an average of 6 months
  The time needed for transition time to total enteral feeding
Daily weight gain | through study completion, an average of 6 months
  The daily weight gain of the infant during the study
Need for anti reflux treatment | through study completion, an average of 6 months
  ıf the infant needed antireflux treatment, the treatment options were recorded
Body weight at discharge | through study completion, an average of 6 months
  Body weight at discharge

CONTACTS AND LOCATIONS:
Overall Officials: Ozge Altun Koroglu, M.D., Study Chair — Ege University
Locations (1):
- Ege University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided